CLINICAL TRIAL: NCT04078919
Title: Effect of Low Calorie Diets With and Without Nuts on Systemic and Vascular Inflammation in Patients With Stable Coronary Artery Disease
Brief Title: Effect of a Low Calorie Diet Containing Nuts on Systemic and Vascular Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Academic Member, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 890
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Diet Therapy; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low calorie diets with nuts (Active Comparator): Low calorie diet in which 20 percent of daily calories will be provided from nuts
  Interventions: Dietary Supplement: Nut consumption; Other: Low calorie diet
- Low calorie diet (Placebo Comparator): Low calorie diet
  Interventions: Other: Low calorie diet

INTERVENTIONS:
Dietary Supplement: Nut consumption — daily consumption of 20 percent of daily calories intake from nuts (pistachio, almond and peanuts)
  Other Names: Dietary Modification
  Arms: Low calorie diets with nuts
Other: Low calorie diet — Low calorie diet

SUMMARY:
Accumulating evidence from prospective observational studies and a large clinical trial suggests that nut intake lowers the risk of cardiovascular disease (CVD). Tree nuts are rich in unsaturated fats, soluble ﬁber, antioxidants, and phytosterols. The purpose of this study is to compare the effects of low calorie diets with a mixture of nuts in comparison with low calorie diets in improving inflammatory markers in patients with stable coronary artery disease.

DETAILED DESCRIPTION:
A randomized placebo controlled clinical trial will be conducted in modares hospital in Tehran, Iran. After review of the inclusion and exclusion criteria and explanation of the design of the study, written consent form will be completed. The participants are 66 eligible patients, aged 35-70 years. Intervention group will be received low calories diets as well as 20 percent of daily calories from mixed nuts (peanuts, pistachio and almond) and control group will be received low calories diets for 8 weeks. Fasting blood sample will be taken to measure inflammatory markers (Interleukine-6 [IL-6] and Interleukine-10 [IL-10] and C-Reactive Protein [CRP]).

ELIGIBILITY:
Inclusion Criteria:

* patients with at least one of the cardiovascular risk factors (hypertension, hyperlipidemia, diabetes mellitus)
* patients with coronary artery disease
* willing to participation in the study

Exclusion Criteria:

* َChronic kidney disease stage 3-5
* Any change in disease treatment plan such as change in type and dose of lipid lowering drugs or surgical operation

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
C reactive protein (CRP) | 8 week
  C reactive protein

SECONDARY OUTCOMES:
inflammatory cytokines | 8 week
  Change in plasma level of inflammatory cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Unit, National Nutrition and Food Technology Research Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghanavati M, Nasrollahzadeh J. A calorie-restricted diet enriched with tree nuts and peanuts reduces the expression of CX3CR1 in peripheral blood mononuclear cells in patients with coronary artery disease. Int J Vitam Nutr Res. 2023 Aug;93(4):329-338. doi: 10.1024/0300-9831/a000738. Epub 2021 Nov 19. PMID 34794330